CLINICAL TRIAL: NCT07117019
Title: Effect of Myofascial Release Combined With Acupressure on BL23 On Chronic Perineal Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Diana Hosny khalil Botros, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005183
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Chronic Perineal Pain
MeSH Terms: interventions — Self Care; Myofascial Release Therapy; Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-care and lifestyle intervention advice (Active Comparator): It will include 20 women suffering from chronic postpartum perineal pain. They will receive self-care and lifestyle intervention advice for four weeks during their daily lifestyle routine.
  Interventions: Other: Self-care and lifestyle intervention advice
- Self-care and lifestyle intervention advice + Myofascial release + Acupressure (Experimental): It will include 20 women suffering from chronic postpartum perineal pain. They will receive the same advice as in the experimental group in addition to myofascial release and acupressure on the BL23 point, three sessions per week for four weeks. The duration of the session will be 40 minutes.
  Interventions: Other: Self-care and lifestyle intervention advice; Other: Myofascial release; Other: Acupressure

INTERVENTIONS:
Other: Self-care and lifestyle intervention advice — All females in both groups will follow self-care and lifestyle advice for 4 weeks.
Other: Myofascial release — Females in the experimental group will receive intravaginal myofascial release in lithotomic position. After ensuring empty bladder/bowel, therapist uses sterile gloves and lubricant to insert fingers 2-3cm into vagina, pressing vaginal walls bilaterally for 2 minutes. Perineal massage follows, targeting scar tissue and tender points with friction at right angles. Treatment duration starts at 5 minutes (due to pain tolerance) and gradually increases to 20 minutes. Hot pack or ultrasound may be used pre-treatment for pain relief. Therapist performs gentle U-shaped reciprocating massage movements up and down towards rectum for 20 minutes total. Sterile technique maintained throughout with hand washing and glove changes between procedures.
  Arms: Self-care and lifestyle intervention advice + Myofascial release + Acupressure
Other: Acupressure — Each female in the experimental group will receive acupressure on BL 23 as follows: Acupressure is also another branch of acupuncture. In this method, fingers press the key points on the skin to stimulate and induce the body's natural self-healing capabilities. In the present study, the BL23 point located 1.5 cm lateral to the lower border of the spinous process of the second lumbar vertebra was employed.
  The therapist will apply pressure on BL 23 points with the thumb for 5 minutes in the counterclockwise direction. In the second 5 minutes, pressure was applied in the opposite direction for 5 minutes. Similarly, the pressure was continued for 20 minutes.
  Arms: Self-care and lifestyle intervention advice + Myofascial release + Acupressure

SUMMARY:
This study aims to determine the effect of the myofascial release combined with acupressure on BL23 on chronic perineal pain.

DETAILED DESCRIPTION:
Perineal pain is a typical sequel vaginal delivery, affecting up to 42% of women at ten days postpartum and persisting in 10% at 18 months. As the fibers of scar tissue form, however, they are typically weaker, with more limited movement and less oxygen circulation than normal skin tissue. This lack of skin and muscle elasticity around an episiotomy or perineal scar can result in side effects, such as pain during sex or when passing a stool, urinary or fecal incontinence, pelvic organ prolapse, and ongoing infections. Moreover, chronic perineal pain can affect the woman psychologically and impact the transition to parenthood, the sexual relationship with her partner, and their ability to breastfeed.

Pharmacological therapies are effective; however, they have side effects as they can pass into breast milk and subsequent harm to the neonate. So, studies need to test and support the effectiveness and safety of some non-pharmacological techniques that could benefit a wide range of women suffering from postpartum perineal pain.

Perineal massage enhances perineal results by stretching the tissues of the vagina, facilitating perineal relaxation, and increasing tissue circulation. Acupressure is a noninvasive method whose nature is similar to acupuncture. This method is effective in sedating pain and reducing its intensity. Some researchers believe that acupressure prevents the transfer of pain stimulators, increases blood endorphin levels, and reduces pain.

Therefore, this study will be carried out to verify the effect of myofascial release and acupressure on postpartum perineal pain.

To our knowledge, this study is the first to investigate the effect of myofascial release combined with acupressure on chronic postpartum perineal pain. Therefore, this study will be conducted to provide physiotherapists with updated scientific knowledge concerning the effect of adding the myofascial release to acupressure on chronic perineal pain, aiming to improve quality of life and decrease pain. This study may expand the role of physiotherapy in women's health.

ELIGIBILITY:
Inclusion Criteria:

1. All women will be diagnosed with chronic perineal pain from episiotomy scar and referred by the gynecologist.
2. Their age will range from 18 to 30 years.
3. They should not have skin irritation/inflammation at the perineum.
4. They should not receive epidural anesthesia, ice packs, or non-steroidal anti-inflammatory drugs during the treatment sessions.
5. They should not suffer from major physical problems such as spinal fractures or disc Hernias.

Exclusion Criteria:

1. Having a laceration other than an episiotomy.
2. Having an operative vaginal delivery (forceps, vacuum).
3. Chronic disease (diabetes mellitus, thyroid, hypertension).
4. Regular medication use or any postnatal complication in the newborn.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-12 (Estimated); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Assessment of intensity of perineal pain | 4 weeks
  The McGill Pain Questionnaire assesses subjective pain experience through three major word descriptor classes: sensory, affective, and evaluative, plus an intensity scale. It provides three quantitative measures: (1) Pain Rating Index (PRI) - based on rank values where words implying least pain=1, increasing sequentially. Separate scores calculated for sensory (subclasses 1-10), affective (11-15), evaluative (16), and miscellaneous (17-20) categories, plus total score (1-20). (2) Number of Words Chosen (NWC) - total descriptors selected. (3) Present Pain Intensity (PPI) - number-word combination indicating overall pain intensity at administration time using 1-5 scale. Designed for statistical analysis of clinical pain.

SECONDARY OUTCOMES:
Assessment of the quality of the scar | 4 weeks
  The Patient and Observer Scar Assessment Scale (POSAS) is a dual-component tool for evaluating scars. The Observer Scale rates 5 variables (vascularity, pigmentation, thickness, relief, pliability, surface area) using 10-point scoring, totaling 5-50 points. The Patient Scale assesses 6 items (pain, itching, color, stiffness, thickness, irregularity) also using 10-point scoring, totaling 6-60 points. Lower scores indicate normal skin. POSAS demonstrates superior internal consistency and inter-observer reliability compared to the Vancouver Scar Scale, with the unique advantage of incorporating patient subjective assessments alongside objective clinical observations, making it ideal for comprehensive post-surgical scar evaluation.
Assessment of quality of life | 4 weeks
  The EuroQol five-dimensional (EQ-5D) is a generic preference-based instrument measuring health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three response levels (1=no problem, 2=moderate problem, 3=severe problem). These can be converted into a summary index score with maximum value of 1 (best health state). Additionally, it includes a visual analogue scale (VAS) rating general health status from 0-100, where 100 represents optimal health. The EQ-5D is widely used for creating health profiles and calculating utility values for economic evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohamed Hanafy, PhD, Study Chair — Professor, Cairo university; Mai Mohamed Ali, PhD, Study Director — Assistant Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt